CLINICAL TRIAL: NCT01694069
Title: Continuous Infusion Piperacillin-Tazobactam for the Treatment of Pulmonary Exacerbations in Patients With Cystic Fibrosis
Brief Title: Continuous Infusion Piperacillin-tazobactam for the Treatment of Cystic Fibrosis
Acronym: PIPE-CF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment was not sufficient to complete the study
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24255
Record Dates: First submitted 2012-09-19; First posted 2012-09-26 (Estimated); Results first posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Cystic Fibrosis
Keywords: piperacillin; tazobactam; pseudomonas aeruginosa; cystic fibrosis; pulmonary exacerbation; continuous infusion; beta lactam
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections | interventions — Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intermittent Infusion piperacillin-tazobactam (Active Comparator): Piperacillin-tazobactam administered at a dose of 400 mg/kg/day (maximum of 16 grams), divided in four equal doses, administered over 30 minutes, four times a day
  Interventions: Drug: Piperacillin-tazobactam combination product
- Continuous infusion piperacillin-tazobactam (Experimental): Piperacillin-tazobactam administered at a dose of 400 mg/kg/day (maximum of 16 grams) as a continuous infusion over 24 hours, once daily
  Interventions: Drug: Piperacillin-tazobactam combination product

INTERVENTIONS:
Drug: Piperacillin-tazobactam combination product — 400 mg/kg/day as either intermittent or continuous infusion
  Other Names: Zosyn

SUMMARY:
Cystic fibrosis is an inherited disorder leading to chronic pulmonary inflammation and infection. A majority of people with cystic fibrosis have large quantities of bacteria residing in their lungs. One of the most common and harmful bacteria is called Pseudomonas aeruginosa.

Patients with cystic fibrosis require frequent therapy with intravenous (I.V.) antibiotics to treat lung infections thought to be caused by Pseudomonas aeruginosa. One of the antibiotics frequently used to treat this bacteria is piperacillin-tazobactam. Piperacillin-tazobactam is thought to be the most effective when there is a constant level of drug in the body. The standard way to administer piperacillin-tazobactam is to give several grams 4 times each day as a 30 minute infusion. An alternative way to give piperacillin-tazobactam is by a continuous infusion; a continuous infusion will make it more likely that drug will remain at a constant level in the body. The objective of this study is to determine if administering piperacillin-tazobactam as a continuous infusion is more effective at treating people having a pulmonary exacerbation of cystic fibrosis than a standard 30 minute infusion, 4 times a day.

DETAILED DESCRIPTION:
All patients will receive combination therapy to include piperacillin-tazobactam 400 mg/kg/day (based on piperacillin component, actual body weight) not to exceed 16 grams and tobramycin 12 mg/kg/day extended interval dosing (once daily). Patients randomized to the continuous infusion group will receive a one-time loading dose of 100 mg/kg over 30 minutes followed immediately by initiation of the continuous infusion.

Other antibiotics with activity against Pseudomonas aeruginosa are not allowed. Patients may receive an antibiotic for treatment of Staphylococcus aureus if deemed appropriate.

Other treatments for pulmonary exacerbation of cystic fibrosis will be left up to the control of the treating physician. Patients will receive a total of 14 days of therapy. If deemed appropriate, patients may be discharged to home where they will continue to receive blinded treatment via an infusion pump. Patients will be evaluated after completing their 14 day course of antibiotics (end of therapy).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cystic fibrosis
2. 8 years of age or greater
3. Chronic or intermittent infection with Pseudomonas aeruginosa as defined by the Leeds Criteria
4. Pulmonary exacerbation as defined by Fuchs et al.

Exclusion Criteria:

1. Admission for greater than 48 hours prior to enrollment
2. Isolation of Burkholderia spp. in a respiratory tract culture in the prior 12 months
3. Current treatment for allergic bronchopulmonary aspergillosis
4. Pregnant or breast feeding
5. History of solid organ transplantation
6. Renal impairment at time of randomization (< 40 mL/min as calculated by the Cockcroft-Gault equation24 ¬for adults or the Schwartz equation45 for those < 18 years of age) or receipt of hemodialysis
7. Allergy to study medication

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Biondo, PharmD, Principal Investigator — West Virginia University Healthcare
Locations (1):
- West Virginia University Healthcare, Morgantown, West Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated and the original PI has left the institution. Minimal results information is available; all efforts were made to retrieve more results information, but were unsuccessful. The available data does not indicate in which arm the participants were enrolled, therefore all available study data with be entered under All Study Participants.
Groups:
- All Study Participants: Intermittent Infusion piperacillin-tazobactam and Continuous infusion piperacillin-tazobactam were combined into the All Study Participants, because the available study data was not separated into arms.
  Continuous infusion piperacillin-tazobactam:
  Piperacillin-tazobactam administered at a dose of 400 mg/kg/day (maximum of 16 grams), divided in four equal doses, administered over 30 minutes, four times a day
  Continuous infusion piperacillin-tazobactam:
  Piperacillin-tazobactam administered at a dose of 400 mg/kg/day (maximum of 16 grams) as a continuous infusion over 24 hours, once daily
  Piperacillin-tazobactam combination product: 400 mg/kg/day as either intermittent or continuous infusion
Period: Overall Study
Arm/Group | All Study Participants
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated and the original PI has left the institution. Minimal results information is available; all efforts were made to retrieve more results information, but were unsuccessful. The available data does not indicate in which arm the participants were enrolled, therefore all available study data with be entered under All Study Participants.
Arm/Group | All Study Participants
Number analyzed (Participants) | 6
Age, Customized [Count of Participants; unit: Participants] — There was no available information about age of participants outside of that included in the inclusion criteria, indicating participants needed to be at least 8 years old to participate.
  Participants
    Between 8 and 99 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Forced Expiratory Volume at One Second (FEV1)
Description: FEV1 will be measured upon enrollment (day 0). FEV1 will also be measured at end of therapy (day 14). If FEV1 is available when patient was stable, prior to enrollment, this value will be treated as baseline FEV1. Change in FEV1 will be calculated from baseline (if available) to day 14 and also Day 0 to day 14
Time Frame: Baseline, Day 0, and Day 14
Population: The study was terminated and the original PI has left the institution. No outcome measure results information is available; all efforts were to made to retrieve results information, but efforts were unsuccessful.
Arm/Group | Intermittent Infusion Piperacillin-tazobactam | Continuous Infusion Piperacillin-tazobactam
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Piperacillin Serum Concentrations
Description: Serum piperacillin concentration will be measured as follows:
  * Intermittent infusion arm: prior to dose (trough), 30 minutes (after completion of infusion), and at 4 hours
  * Continuous infusion arm: collected at the same time as in the intermittent infusion arm
Time Frame: Day 3
Population: as for outcome 1
Arm/Group | Intermittent Infusion Piperacillin-tazobactam | Continuous Infusion Piperacillin-tazobactam
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Next Pulmonary Exacerbation
Description: Patients will be followed for time of next subsequent pulmonary exacerbation for up to 52 weeks after completion of receiving study drug. Next pulmonary exacerbation is defined as requiring admission to a hospital for receipt of I.V. antibiotics because of a diagnosis of pulmonary exacerbation.
Time Frame: Patients will be followed up to 52 weeks from time of enrollment
Population: as for outcome 1
Arm/Group | Intermittent Infusion Piperacillin-tazobactam | Continuous Infusion Piperacillin-tazobactam
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Score
Description: The validated CFQ-R will be administered to patients at time of enrollment at end of therapy
Time Frame: Day 0 and day 14
Population: as for outcome 1
Arm/Group | Intermittent Infusion Piperacillin-tazobactam | Continuous Infusion Piperacillin-tazobactam
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Sputum Density of Pseudomonas Aeruginosa
Description: Sputum density of Pseudomonas aeruginosa will be determined at enrollment, day 3, and at end of therapy
Time Frame: Day 0, day 3, and day 14
Population: as for outcome 1
Arm/Group | Intermittent Infusion Piperacillin-tazobactam | Continuous Infusion Piperacillin-tazobactam
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Weight
Description: The change in weight will be documented from enrollment to end of therapy
Time Frame: Day 0 and day 14
Population: as for outcome 1
Arm/Group | Intermittent Infusion Piperacillin-tazobactam | Continuous Infusion Piperacillin-tazobactam
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Time to Defervescence
Description: Temperature will be taken multiple times daily according to standard of care. If patients present febrile, time until patient is afebrile and remains afebrile for 24 hours will be recorded.
Time Frame: Day 0 to day 14
Population: as for outcome 1
Arm/Group | Intermittent Infusion Piperacillin-tazobactam | Continuous Infusion Piperacillin-tazobactam
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Time to Normalization of White Blood Cell Count
Description: White blood cell (WBC) count will be measured once daily. If patient presents with WBC count greater than 11.0 x 10^3/mL, time until patient has WBC less than 11.0 x 10^3/mL will be recorded.
Time Frame: Day to day 14
Population: as for outcome 1
Arm/Group | Intermittent Infusion Piperacillin-tazobactam | Continuous Infusion Piperacillin-tazobactam
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Clinical Failure of Treatment
Description: Failure of treatment will be defined as patient needing I.V. antibiotics beyond the 14 days allowed in this study. The primary medical team (along with a blinded investigator) treating the patient will determine whether patient requires additional therapy.
Time Frame: Day 14
Population: as for outcome 1
Arm/Group | Intermittent Infusion Piperacillin-tazobactam | Continuous Infusion Piperacillin-tazobactam
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The study was terminated and the original PI has left the institution. No adverse event information is available; all efforts were to made to retrieve adverse event information, but efforts were unsuccessful.
Arm/Group | Intermittent Infusion Piperacillin-tazobactam | Continuous Infusion Piperacillin-tazobactam
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes